CLINICAL TRIAL: NCT00397761
Title: Combination Capecitabine (Xeloda) and ABI-007 (Abraxane, Nanoparticle Albumin-Bound Paclitaxel) Chemotherapy as Neoadjuvant Treatment of Locally Advanced, Operable Breast Cancer
Brief Title: Capecitabine and Paclitaxel (Albumin-Stabilized Nanoparticle Formulation) in Treating Women Undergoing Surgery for Stage II or Stage III Breast Cancer
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000513169; WHC-MRI-GU-2006-097
Record Dates: First submitted 2006-11-08; First posted 2006-11-09 (Estimated); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Breast Cancer
Keywords: inflammatory breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer
MeSH Terms: conditions — Breast Neoplasms; Inflammatory Breast Neoplasms | interventions — Capecitabine; Taxes; Neoadjuvant Therapy

INTERVENTIONS:
Drug: capecitabine
Drug: paclitaxel albumin-stabilized nanoparticle formulation
Procedure: neoadjuvant therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as capecitabine and paclitaxel (albumin-stablized nanoparticle formulation, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

PURPOSE: This phase II/III trial is studying how well giving capecitabine together with paclitaxel (albumin-stabilized nanoparticle formulation) works in treating women undergoing surgery for stage II or stage III breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the rate of pathological complete response (i.e., tumor completely gone) in women with previously untreated, unresected, stage II-IIIB breast cancer treated with neoadjuvant therapy comprising capecitabine and paclitaxel (albumin-stabilized nanoparticle formulation) (Abraxane^®).

Secondary

* Evaluate the safety of this regimen in these patients.
* Determine overall clinical response rate in patients treated with this regimen.

OUTLINE: Patients receive up to 4 courses of capecitabine and paclitaxel (nanoparticle albumin-stabilized formulation) (Abraxane^®) in the absence of disease progression. Patients then undergo definitive surgical resection of the tumor off study.

PROJECTED ACCRUAL: A total of 33 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed infiltrating carcinoma of the breast or inflammatory breast cancer

  * Stage II-IIIB disease (T1-4, N1-2, M0)
* Previously untreated disease
* Previously unresected disease
* High-risk disease that is not resectable by lumpectomy alone
* Any HER2/neu status (positive, negative, or unknown) allowed
* Hormone receptor status:

  * Any estrogen/progesterone status (positive, negative, or unknown) allowed

PATIENT CHARACTERISTICS:

* Female
* Menopausal status not specified
* ECOG performance status 0-2
* Life expectancy > 3 months
* Absolute neutrophil count > 1,500/mm³
* Platelet count > 100,000/mm³
* Hemoglobin > 9.0 g/dL
* Creatinine < 1.5 mg/dL
* Bilirubin < 1.5 times upper limit of normal (ULN)
* ALT and AST < 2.5 times ULN (5 times ULN if due to Gilbert's disease)
* Alkaline phosphatase < 2.5 times ULN (5 times ULN if due to Gilbert's disease)

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-07

PRIMARY OUTCOMES:
Pathological complete response rate

SECONDARY OUTCOMES:
Safety
Overall clinical response rate

CONTACTS AND LOCATIONS:
Overall Officials: Anita Aggarwal, DO, PhD, Study Chair — Medstar Health Research Institute
Locations (1):
- Washington Cancer Institute at Washington Hospital Center, Washington D.C., District of Columbia, United States